CLINICAL TRIAL: NCT03344575
Title: Randomised Controlled Trial of Peritoneal Bridging Versus Defect Closure in Laparoscopic Ventral Hernia Repair
Brief Title: Peritoneal Bridging in Laparoscopic Ventral Hernia Repair
Acronym: BriClo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karlskoga Hospital (Unknown)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BriClo
Record Dates: First submitted 2017-11-12; First posted 2017-11-17 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Hernia, Ventral; Laparoscopy; Seroma
MeSH Terms: conditions — Hernia, Ventral; Seroma

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient undergoing surgery and the physician performing the follow-up are masked to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional defect closure (Active Comparator): The defect is sutured with continuous PDS 2-0.
  Interventions: Procedure: Conventional defect closure
- Peritoneal bridging (Experimental): The peritoneum is dissected beginning 2-3 cm from the edge of the defect. The sac is dissected all the way to the opposite edge of the defect. The peritoneal flap is pulled to the opposite side and fixated with Optifix
  Interventions: Procedure: Peritoneal bridging

INTERVENTIONS:
Procedure: Conventional defect closure — Laparoscopic suturing of the defect prior to placing an intraperitoneal Onlay Mesh
  Arms: Conventional defect closure
Procedure: Peritoneal bridging — Laparoscopic closure of the defect by using a peritoneal flap prior to placing an intraperitoneal Onlay Mesh
  Arms: Peritoneal bridging

SUMMARY:
Laparoscopic ventral hernia repair (VHR) is usually performed by reducing the contents in the hernia sac from the abdominal cavity and then covering the defect from the inside with a mesh, i.e. Intraperitoneal Onlay Mesh (IPOM). This means that the hernia sac is left in situ anterior to the mesh. This may, however, predispose for the development of fluid in the hernia sac, i.e. seroma. The risk of seroma development may be reduced if a the defect is closed before the mesh is applied. Closing the defect may, however, cause tension and pain from the abdominal wall. Instead of closing the defect, the part of the peritoneum constituting the hernia sac may be used for closing the defect. In this case, the peritoneum is dissected from the edges of the hernia sac and then used as a flap that is fixated to the edges of the hernia sac on the opposite side.

In order to evaluate whether peritoneal bridging reduces the seroma development following ventral hernia repair, we are undertaking a double-blind randomized controlled trial comparing conventional closure of the hernia defect with peritoneal bridging. The goal is to randomize 50 patients undergoing laparoscopic ventral hernia to conventional closure or closure of the defect with peritoneal bridging.

Clinical follow-up is performed one month and one year after surgery. At both occasions, the patient is requested to fill in the Ventral Hernia Pain Questionnaire (VHPQ) and an investigation is done in order to assess the presence of seromas, recurrences or other local complications. One year after surgery, computer tomography is performed. The main purpose of the computer tomography is to quantify the presence of seromas.

The study is intended as phase 2 study with the aim of evaluating peritoneal bridging as an alternative to conventional defect closure. If the study shows that bridging does not lead to substantial seroma development, future studies with greater statistical power and other outcome measures will be undertaken.

DETAILED DESCRIPTION:
Background

Laparoscopic ventral hernia repair (VHR) has become a well-established technique during the last decade. The repair is usually performed by reducing the contents in the hernia sac from the abdominal cavity and then covering the defect from the inside with a mesh, i.e. Intraperitoneal Onlay Mesh (IPOM). This means that the hernia sac is left in situ anterior to the mesh. This may, however, predispose for the development of fluid in the hernia sac, i.e. seroma. Even if the mesh prevents the intestines from protruding into the hernia sac, the patient may still be troubled by discomfort from the seroma that replaces the hernia..

The risk of seroma development may be reduced if a the defect is closed before the mesh is applied (IPOM-Plus). Closing the defect may, however, cause tension and pain from the abdominal wall. Instead of closing the defect, the part of the peritoneum constituting the hernia sac may be used for closing the defect. In this case, the peritoneum is dissected from the edges of the hernia sac and then used as a flap that is fixated to the edges of the hernia sac on the opposite side. This reduces the size of the pseudosac and the peritoneal surface, which prevents transudation to the pseudosac.

In order to evaluate whether peritoneal bridging reduces the seroma development following ventral hernia repair, we are undertaking a randomized controlled trial. Our goal is to include 50 patients in the study.

Method

After obtaining written and oral consent from the patient, the randomisation is performed through a sealed envelope system. The patient is blinded to the allocation. Prior to the procedure, the patient is also requested to fill in the Ventral Hernia Pain Questionnaire (VHPQ).

The procedure is started according to the usual routines. Adhesions covering the defect are dissected in order to visualize the defect. If the patients has been randomized to defect closure, it is sutured with continuous PDS 2-0. . In case the patient is allocated to peritoneal bridging, the peritoneum is dissected beginning 2-3 cm from the edge of the defect. The sac is disected all the way to the opposite edge of the defect. The peritoneal flap is pulled to the opposite side and fixated with Optifix. One of the aims of the bridging is to to close the defect and increase the surface of contact between the mesh and the peritoneum.

The mesh is attached in the same, irrespective of randomization. Optifix with double-crown technique is used in both groups. Operation time and intraoperative complications are registered when the procedure is completed. From the day of the procedure until two days postoperatively, pain from the area of surgery is registered daily on a VAS-scale.

The patient is invited to clinical follow-up one month and one year after surgery. At both occasions the patient is requested to fill in VHPQ. One year after surgery, a computer tomography while straining in order to detect protrusion of the abdominal contents in the defect. Any protrusion seen at the computer tomography is graded according to a previously validated classification. The presence of seromas detected at the computer tomography is described according to Morales-Conde,

The computer tomography images are assessed by two radiologists in order to reach consensus. The presence of seroma anterior to the defect is evaluated in terms of size (maximal diameter), localization, shape (round, oval, triangular), mean density (Hounsfield unit, HU) and the volume through three-dimensional reconstructions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients planned for laparoscopic repair of midline incisional hernia
* Defects with diameter 3-10 cm
* BMI<40

Exclusion Criteria:

* Defect >10 cm
* Ventral hernias with other localization than the midline
* Emergency surgery and incarcerated hernias
* Preoperative suspicion of extensive adhesions
* Pregnancy or intended pregnancy
* Serious comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Seroma formation | One year
  Volume of postoperative seroma measured with computer tomography

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  Complications related to the procedure
Postoperative pain | One year
  Pain assessed with the Ventral Hernia Pain Questionnaire for rating abdominal wall pain. Range 0-7 from no pain to most intensive pain. No subscales or added scores.
Time required to close the defect | 3 hours
  Time (minutes) from beginning the closure to placing the mesh
Hernia recurrence | One year
  Recurrence of the hernia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Karloskoga Hospital, Karlskoga, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali F, Wallin G, Fathalla B, Sandblom G. Peritoneal bridging versus fascial closure in laparoscopic intraperitoneal onlay ventral hernia mesh repair: a randomized clinical trial. BJS Open. 2020 Aug;4(4):587-592. doi: 10.1002/bjs5.50305. Epub 2020 May 28. PMID 32463163